CLINICAL TRIAL: NCT06283121
Title: A Clinical Study to Evaluate the Safety and Efficacy of Recombinant Human nsIL12 Oncolytic Adenovirus Injection (BioTTT001) in Combination With SOX and Toripalimab in Patients With Peritoneal Metastases From Gastric Cancer
Brief Title: A Clinical Study of BioTTT001 in Combination With SOX and Toripalimab in Patients With Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University, China (Other)
Collaborators: Beijing Bio-Targeting Therapeutics Technology Co., Ltd (Industry)
Responsible Party: Principal Investigator, Funan Liu, professor, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJCT-CMU1H-01
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer, Metastatic
Keywords: oncolytic virus; IL-12; gastric cancer; peritoneal metastases
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination therapy with BioTTT001 intraperitoneal infusion , SOX and Toripalimab (Experimental): This study intends to enroll Her2-negative subjects with first-line treatment of peritoneal metastasis from gastric cancer. Subjects will be treated with BioTTT001 intraperitoneal perfusion combined with SOX and toripalimab after completing the screening period, and the subjects will first receive BioTTT001 monotherapy treatment with BioTTT001 1×10^10 VP intraperitoneal perfusion (P.I.), D1 and D3, and enter the combination therapy stage 7 days (±1d) after the first dose of BioTTT001.Subjects will be treated with the regimen as follows: BioTTT001 injection, 1×10^10 VP P.I., D1；toripalimab 160mg intravenous (i.v.), D1; Oxaliplatin 130mg/m^2 i.v. , D1 ; Tegafur 40~60mg Bis in die（b.i.d.） Peroral（p.o.）D1~D14; 3 weeks per cycle.
  Interventions: Biological: BioTTT001 intraperitoneal infusion; Drug: SOX regimen; Drug: toripalimab

INTERVENTIONS:
Biological: BioTTT001 intraperitoneal infusion — Monotherapy lead-in phase: BioTTT01 1×10^10 VP, i.p., D1 and D3; Combination therapy phase: BioTTT01 1×10^10 VP, i.p., D1 and D3, 3 weeks per cycle
Drug: SOX regimen — Combination therapy phase: Oxaliplatin 130 mg，i.v., D1 and D3, 3 weeks per cycle; Tegafur 40~60mg b.i.d. p.o. D1~D14; 3 weeks per cycle
Drug: toripalimab — Combination therapy phase: toripalimab 160mg i.v. D1, 3 weeks per cycle.

SUMMARY:
This is a phase I, single arm, open-label clinical study of BioTTT001 in combination with SOX and Toraplizumab in patients with peritoneal metastases from gastric cancer.

DETAILED DESCRIPTION:
This study intends to enroll Her2-negative subjects with first-line treatment of peritoneal metastasis from gastric cancer. Subjects will be treated with BioTTT001 intraperitoneal perfusion combined with SOX and toripalimab after completing the screening period, and the subjects will first receive BioTTT001 monotherapy treatment with BioTTT001 1×10^10 viral particle (VP) intraperitoneal perfusion (P.I.), D1 and D3, and enter the combination therapy stage 7 days (±1d) after the first dose of BioTTT001.Subjects will be treated with the regimen as follows: BioTTT001 injection, 1×10^10 VP P.I., D1；toripalimab 160mg intravenous (i.v.), D1; Oxaliplatin 130mg/m^2 i.v. , D1 ; Tegafur 40~60mg Bis in die（b.i.d.） Peroral（p.o.）D1~D14; 3 weeks per cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age≥ 18 years；
2. Patients with a diagnosis of gastric cancer by histopathology or cytology, accompanied by peritoneal metastasis, without systemic therapy, or for patients who have received neoadjuvant/adjuvant chemotherapy before, the time from last treatment to disease recurrence > 6 months;
3. Tumor Her2 negative (IHC 0/1＋ or IHC 2＋ and FISH-).
4. At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors （RECIST) 1.1;
5. WBC≥3.0×10^9 /L; ANC≥1.5×10^9 /L; HB≥90 g/L; PLT≥75×10^9 /L;
6. ALT and AST≤3×ULN (≤5×ULN with liver metastasis); ALB≥20g/L; Cr≤1.5×ULN or CCr>50 mL/min; TBIL≤1.5×ULN; APTT≤1.5×ULN and INR or PT≤1.5×ULN (without anticoagulation therapy)
7. LVEF≥50%; male QTc≤450 mms, female QTc≤470 mms;
8. ECOG 0~1；
9. Expected survival ≥ 3 months;
10. Consent to contraception；
11. Understand and voluntarily sign a written ICF and be willing to comply with all trial requirements.

Exclusion Criteria:

1. History of other malignancies (except cured basal cell skin cancer, cervical carcinoma in situ etc.) within 5 years before study drug administration;
2. Patients with central nervous system metastases with clinical symptoms;
3. Patients who have been treated with high-dose systemic corticosteroids (prednisone > 10 mg/day or equivalent doses) or other immunosuppressants within 2 weeks before the first dose of BioTTT001;
4. Previous treatment with other adenovirus drugs within 28 days before the first dose of BioTTT001;
5. Patients who have undergone any major surgery (except needle biopsy, etc.) or severe trauma within 14 days before the first dose of BioTTT001;
6. Patients who have not recovered from the adverse reactions of previous treatments (the treatment-related toxicity ≤ grade 2, except for alopecia );
7. Patients with primary immunodeficiency;
8. Patients with active autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, etc.), except type 1 diabetes, hypothyroidism that only needs hormone replacement therapy, and skin diseases that do not need systemic treatment (such as vitiligo, psoriasis or alopecia);
9. Patients with active infection requiring systemic anti-infective therapy;
10. HBsAg positive, and blood HBV DNA≥100 IU/mL; anti-HCV positive; HIV positive; active syphilis;
11. Patients with active tuberculosis or drug-induced interstitial lung disease；
12. Patients with active inflammatory bowel disease ；
13. NYHA≥ grade 3；
14. Known allergy to the investigational drug or its components;
15. Patients with prior organ transplants;
16. Pregnant or lactating women;
17. Other reasons judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-02 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Imaging was performed every 6 weeks during the combination therapy phase
  Objective response rate (ORR) as assessed by the investigators

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Every 6 weeks until disease progression, consent withdraw, death or end of study during the combination therapy phase, up to 100 weeks.
  The time from the start of treatment to progress disease or death for any cause
Overall survival (OS) | Every 3 months until consent withdraw, death, withdrawal study, or loss of follow-up, up to 100 weeks
  The time from the start of treatment to death for any cause

CONTACTS AND LOCATIONS:
Overall Officials: Zhenning Wang, MD, Principal Investigator — The First Affiliated Hospital of China Medical Univeristy; Funan Liu, MD, Principal Investigator — The First Affiliated Hospital of China Medical Univeristy